CLINICAL TRIAL: NCT05203822
Title: Phase I, Open-label, Single-sequence, Cross-over Study of the Effect of Multiple Doses of Itraconazole on Single-dose Tepotinib Pharmacokinetics in Healthy Participants
Brief Title: Tepotinib Drug-Drug Interaction Study With Itraconazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200095_0053; 2021-003513-19 (EudraCT Number)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Clinical pharmacology; Metabolite; Induction of metabolism
MeSH Terms: interventions — tepotinib; Itraconazole

STUDY DESIGN:
Intervention Model Description: This is a single sequence cross-over trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tepotinib then Itraconazole (Experimental): Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day and Day 12 under fed condition followed by single oral dose of itraconazole 200 mg on Days 8 to 11 and Days 13 to 18. On Day 12, participants received a single dose of 200 mg itraconazole simultaneously with a single dose of 500 mg Tepotinib.
  Interventions: Drug: Tepotinib (HydroChloride hydrate); Drug: Itraconazole

INTERVENTIONS:
Drug: Tepotinib (HydroChloride hydrate) — Participants received Tepotinib (Hydrochloride hydrate) Film-coated tablet with food on Day 1 and 12 in the morning.
Drug: Itraconazole — Participants received Itraconazole Hard-gelatin capsule with food once daily at the same time in the morning from Day 8 to Day 18; on Day 12 itraconazole is administered concomitantly with tepotinib.

SUMMARY:
The purpose of this study was to assess the effect of multiple doses of itraconazole on single dose tepotinib pharmacokinetics in healthy participants. Study details include:

Study Duration: up to 48 days Treatment Duration: single dose of tepotinib on Days 1 and 12, 11 days of treatment with itraconazole (Days 8 to 18) Visit Frequency: residence in the Clinical Research Unit from Days -1 to 4 and Days 11 to 15, ambulatory daily visits from Days 5 to 10 and 16 to 20

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants as determined by medical evaluation, including no clinically significant abnormality identified by medical history, cardiac monitoring, physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion at Screening and Day -1
* Had a body weight within 50 and 100 kilogram (inclusive) and Body Mass Index (BMI) within the range greater than or equal (>=) 18.5 and less than or equal to (<=) 29.9 kilogram per meter square (inclusive) at Screening
* Male or female (not a Women of childbearing potential [WOCBP]). The Investigator confirms that each participant agrees to use appropriate contraception and barriers, if applicable. The contraception, barrier, and pregnancy testing requirements are below:
* Contraceptive use will be consistent with local regulations on contraception methods for those participating in clinical studies. Male Participants: Agree to the following during the study intervention period and for at least 1 week after the last dose of study intervention: Refrain from donating fresh and unwashed sperm PLUS, either: Abstain from intercourse with a WOCBP.OR Use a male condom: When having sexual intercourse with a WOCBP, who is not currently pregnant, and instruct her to use a highly effective contraceptive method with a failure rate of < 1percent (%) per year
* Not a WOCBP, confirmed at Screening, by fulfilling at least 1 of the following criteria: Females who are postmenopausal and documentation of irreversible surgical sterilization by hysterectomy, or bilateral oophorectomy, or bilateral salpingectomy
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and this protocol
* All values for hematology, coagulation, and biochemistry tests of blood and urinalysis within the normal range (at Screening and Day -1)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Participants with gall bladder removal or other relevant surgery of gastrointestinal tract (appendectomy is not considered as relevant)
* History of any malignancy except for adequately treated superficial basal cell carcinoma
* History of epilepsy
* Ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or excipients; history of anaphylaxis to drugs or serious allergic reactions leading to hospitalization or any other allergy reaction in general, which the Investigator considers may affect the safety of the participant and/or outcome of the study
* Any condition, including findings in the laboratory tests, medical history, or other Screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Use of any prescribed medicine or over-the-counter drug or dietary supplement, including herbal remedies, vitamins, and minerals, antacids and dietary supplements such as fish oils within 2 weeks or 5 times the half-life of the respective drug, whichever is longer, prior to the first administration of study intervention
* Participation in the treatment phase of a clinical study within 60 days or 5 half-lives after last dosing of the previous study drug, whatever is longer, before administration of study drug
* Contraindication to itraconazole: ventricular dysfunction such as congestive heart failure or a history of congestive heart failure, drug interactions (example: co-administration of a number of CYP3A4 substrates), pregnancy, hypersensitivity to itraconazole
* Donation or loss of more than 450 milliliter (mL) of blood in the 60 days prior to Screening, donation of plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening
* Consumption of alcohol from 48 hours prior to first administration of study intervention
* Smoker (cigarettes, pipes, cigars, or others) or former smoker who stopped smoking for less than 6 months before the time of the Screening visit
* Inability to communicate or cooperate with the Investigator (example: language problem, illiteracy, poor mental status) or to comply with the requirements of the entire study, including dietary restrictions
* Other factors, which in the opinion of the Investigator may interfere with study conduct
* Legal incapacity or limited legal capacity
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 participants were screened, out of which 18 participants received the study drug.
Groups:
- Tepotinib and Itraconazole: Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 1 and Day 12 under fed condition followed by single oral dose of itraconazole 200 mg on Days 8 to 11 and Days 13 to 18. On Day 12, participants received a single dose of 200 mg itraconazole simultaneously with a single dose of 500 mg tepotinib.
Period: Overall Study
Arm/Group | Tepotinib and Itraconazole
Started | 18
Completed | 16
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) included all participants, who were administered any dose of any study intervention.
Arm/Group | Tepotinib and Itraconazole
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Tepotinib
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda (λ)z determination.
Time Frame: Predose up to 168 hours post dose
Population: Pharmacokinetic (PK) analysis set included all participants who were administered any dose of any study intervention and completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* nanograms per milliliter(h*ng/mL)
Groups:
- Tepotinib: Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 1.
- Tepotinib and Itraconazole: Participants received 200 mg itraconazole with food once daily in the morning from Day 12 to Day 18 along with a single oral dose of Tepotinib 500 mg on Day 12.
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
hours* nanograms per milliliter(h*ng/mL) | 18927 (28.2) | 23158 (29.9)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Time of Last Measurable Concentration (AUC0-tlast) of Tepotinib
Description: The AUC from time zero (= dosing time) to time of the last quantifiable concentration (tlast). Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Predose up to 168 hours post dose
Population: PK analysis set included all participants who were administered any dose of any study intervention and completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Tepotinib: Participants received a single oral dose of Tepotinib 500 mg on Day 1.
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
h*ng/mL | 18300 (27.9) | 21391 (30.2)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib and Metabolite
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Predose up to 168 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter (ng/mL)
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
nanogram per mililiter (ng/mL) | 308 (24.8) | 313 (28.2)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAES With Severity of Grade Greater or Equal to 3
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE's were those events with onset dates on or after the first administration of study intervention. Severity of abnormalities were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version [24.1].
  grade 1 : mild grade 2 : moderate grade 3 : severe or medically significant but not immediately life-threatening grade 4 : life threatening or disabling grade 5 : death related to AE
Time Frame: Baseline (Day 1) up to follow up (assessed up to Day 20)
Population: The Safety Analysis Set (SAF) included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib and Itraconazole
Number analyzed (Participants) | 18
Participants
  Any TEAE | 14
  Any serious TEAE | 0
  Any TEAE of Grade ≥ 3 (severe) | 0

5. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Laboratory Values
Description: Laboratory investigation included hematology, biochemistry and urinalysis. Clinically meaningful was decided by the investigator. Number of participants with clinically meaningful change from baseline in laboratory values were reported.
Time Frame: Baseline (Day 1) up to follow up (assessed up to Day 20)
Population: SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib and Itraconazole
Number analyzed (Participants) | 18
Participants
  Hematology | 0
  Biochemistry | 0
  Urinalysis | 0

6. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG)
Description: The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT and QTcB calculated by the Bazett formula. Clinical Significance was decided by the investigator. Number of participants with clinically meaningful change from baseline in ECG parameters were reported.
Time Frame: Baseline (Day 1) up to follow up (assessed up to Day 20)
Population: SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib and Itraconazole
Number analyzed (Participants) | 18
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs
Description: Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. Clinical Significance was decided by the investigator. Number of participants with clinically significant change from baseline in vital signs.
Time Frame: Baseline (Day 1) up to follow up (assessed up to Day 20)
Population: SAF included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib and Itraconazole
Number analyzed (Participants) | 18
Participants | 0

8. Secondary Outcome: Total Body Clearance of Drug From Plasma (CL/f) for Tepotinib
Description: CL/f following oral administration was calculated as Dose/AUC0-inf, where AUC0-inf calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastcalc/λz, where Clastcalc was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and λz was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Predose up to 168 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
liter/hour | 23.8 (28.2) | 19.4 (29.9)

9. Secondary Outcome: Apparent Volume of Distribution (Vz/f) for Tepotinib
Description: Vz/F was defined as the apparent volume of distribution during the terminal phase following extravascular administration.
Time Frame: Predose up to 168 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
liters | 1102 (29.4) | 1148 (34.3)

10. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib
Description: The time to reach the maximum observed plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Predose up to 168 hours post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
hours | 8.00 [6.00 to 16.00] | 8.00 [6.05 to 24.00]

11. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Tepotinib in Plasma
Description: t1/2 was defined as the time taken for the plasma concentration or the amount of drug in the body to be reduced by half.
Time Frame: Predose up to 168 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tepotinib | Tepotinib and Itraconazole
Number analyzed (Participants) | 17 | 17
hours | 32.1 (7.8) | 40.9 (19.2)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to follow up (assessed up to Day 20)
Arm/Group | Tepotinib and Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 14/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tepotinib and Itraconazole (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Faeces hard (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1
Catheter site induration (General disorders) | 1
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 2
Rhinitis (Infections and infestations) | 1 (1)
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Clumsiness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Abnormal dreams (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 4
Nocturia (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT05203822/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT05203822/SAP_001.pdf